CLINICAL TRIAL: NCT02441361
Title: Effects of Exercise in Bariatric Patients: a Randomized Controlled Trial
Brief Title: Effects of Exercise Training in Bariatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise & Bariatric
Record Dates: First submitted 2015-03-31; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Subjects will undergo bariatric surgery and no exercise training will be prescribed.
- exercise training (Experimental): Subjects will undergo bariatric surgery and exercise training will be prescribed.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Exercise training will comprise aerobic and strength exercises
  Arms: exercise training

SUMMARY:
Bariatric surgery may attenuate insulin resistance and low-grade inflammation in obese subjects. This trial aims to test whether exercise training can add to the benefits of bariatric surgery on insulin sensitivity and inflammation. In addition, this study aims to investigate whether exercise training can counteract bone loss induced by bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 35 kg/m2
* not engaged in physical activity programs
* without any physical limitation that could preclude exercise participation

Exclusion Criteria:

* body mass index < 35 kg/m2
* regular participation in physical activities programs
* cancer or any other disease that could limit participation in exercise

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity as assessed by surrogates of insulin sensitivity | 6 months
body composition as assessed by densitometry (DEXA) | 6 months
  bone mass, lean mass and fat mass
profile of cytokines | 6 months

SECONDARY OUTCOMES:
physical activity level as assessed by accelerometry | 6 months
quality of life as assessed by questionnaires (composite) | 6 months
muscle function as assessed by a battery of tests | 6 months
  timed-stands test, timed-up-ang-go test, maximal strength tests
risk of cardiovascular events as assessed by questionnaires (composite) | 6 months
aerobic conditioning as assessed by a cardiopulmonary test. | 6 months
depression and anxiety as assessed by questionnaires (composite) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Merege-Filho CAA, Gil SS, Kirwan JP, Murai IH, Dantas WS, Nucci MP, Pastorello B, de Lima AP, Bazan PR, Pereira RMR, de Sa-Pinto AL, Lima FR, Brucki SMD, de Cleva R, Santo MA, Leite CDC, Otaduy MCG, Roschel H, Gualano B. Exercise modifies hypothalamic connectivity and brain functional networks in women after bariatric surgery: a randomized clinical trial. Int J Obes (Lond). 2023 Mar;47(3):165-174. doi: 10.1038/s41366-022-01251-8. Epub 2022 Dec 30. PMID 36585494
- [Derived] Gil S, Kirwan JP, Murai IH, Dantas WS, Merege-Filho CAA, Ghosh S, Shinjo SK, Pereira RMR, Teodoro WR, Felau SM, Benatti FB, de Sa-Pinto AL, Lima F, de Cleva R, Santo MA, Gualano B, Roschel H. A randomized clinical trial on the effects of exercise on muscle remodelling following bariatric surgery. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1440-1455. doi: 10.1002/jcsm.12815. Epub 2021 Oct 19. PMID 34666419
- [Derived] Dantas WS, Roschel H, Murai IH, Gil S, Davuluri G, Axelrod CL, Ghosh S, Newman SS, Zhang H, Shinjo SK, das Neves W, Merege-Filho C, Teodoro WR, Capelozzi VL, Pereira RM, Benatti FB, de Sa-Pinto AL, de Cleva R, Santo MA, Kirwan JP, Gualano B. Exercise-Induced Increases in Insulin Sensitivity After Bariatric Surgery Are Mediated By Muscle Extracellular Matrix Remodeling. Diabetes. 2020 Aug;69(8):1675-1691. doi: 10.2337/db19-1180. Epub 2020 May 14. PMID 32409493
- [Derived] Murai IH, Roschel H, Dantas WS, Gil S, Merege-Filho C, de Cleva R, de Sa-Pinto AL, Lima F, Santo MA, Benatti FB, Kirwan JP, Pereira RM, Gualano B. Exercise Mitigates Bone Loss in Women With Severe Obesity After Roux-en-Y Gastric Bypass: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4639-4650. doi: 10.1210/jc.2019-00074. PMID 31322672